CLINICAL TRIAL: NCT03429153
Title: Impact of Setting up a Multidisciplinary Consensus Meeting in the Prognosis and Management of Infectious Endocarditis at Strasbourg University Hospital.
Brief Title: Management of Infectious Endocarditis as Part of a Multidisciplinary Consensus Meeting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6817
Record Dates: First submitted 2018-01-05; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-01

CONDITIONS: Endocarditis
Keywords: endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
New ESC 2015 recommendations with encouragement to set up a Multidisciplinary Consultation Meeting to discuss the medical and surgical management of endocarditis, set up at Strasbourg University Hospital in October 2016: Impact and benefits

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 18 years at diagnosis
* Diagnosis of confirmed Infectious Endocarditis
* Medical and / or surgical care at Strasbourg University Hospital between January 2007 and June 2018

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Diagnosis of confirmed Infectious Endocarditis
  * Medical and / or surgical care at Strasbourg University Hospital between January 2007 and June 2018
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xavier ARGEMI, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de Maladies Infectieuses et Tropicales, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No